CLINICAL TRIAL: NCT02592486
Title: A Randomized, Open-label, Parallel Design Study to Compare the Immunogenicity of Simultaneous Administration Versus Sequential Administration of Quadrivalent Influenza Vaccine and 23-valent Pneumococcal Vaccine
Brief Title: The Immunogenicity of Simultaneous Administration of Quadrivalent Influenza Vaccine and 23-valent Pneumococcal Vaccine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kameda Medical Center (Other)
Collaborators: PPD Development, LP (Industry); Osaka University (Other); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Kei Nakashima, Assistant Chief, Department of Pulmonary Medicine, Kameda Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 15-041-160127
Record Dates: First submitted 2015-10-28; First posted 2015-10-30 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Pneumococcal Pneumonia; Influenza
Keywords: quadrivalent influenza vaccine; 23-valent pneumococcal vaccine; immunogenicity
MeSH Terms: conditions — Pneumonia, Pneumococcal; Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Simultaneous administration group (Active Comparator): The subjects receive injections of pneumococcal vaccine and influenza vaccine simultaneously. We use commercially available PPV23 (Pneumovax NP®, MSDKK, Tokyo, Japan) containing 25 μg each of 23 capsular polysaccharide types. We use Fluvic HA syringe® (Handai Biken Ltd, Osaka, Japan), quadrivalent influenza vaccine (0.5ml) of 2015/2016 season.
  Interventions: Biological: Simultaneous administration of Pneumovax NP® and Fluvic HA syringe®
- Sequential administration group (Active Comparator): The subjects receive injections of pneumococcal vaccine 2 weeks after the injection of the influenza vaccine. We use commercially available PPV23 (Pneumovax NP®, MSDKK, Tokyo, Japan) containing 25 μg each of 23 capsular polysaccharide types. We use Fluvic HA syringe® (Handai Biken Ltd, Osaka, Japan), quadrivalent influenza vaccine (0.5ml) of 2015/2016.
  Interventions: Biological: Sequential administration of Pneumovax NP® and Fluvic HA syringe®

INTERVENTIONS:
Biological: Simultaneous administration of Pneumovax NP® and Fluvic HA syringe® — Injections of pneumococcal vaccine and influenza vaccine simultaneously.
  Other Names: Pneumovax NP® and Fluvic HA syringe®
  Arms: Simultaneous administration group
Biological: Sequential administration of Pneumovax NP® and Fluvic HA syringe® — Injections of pneumococcal vaccine 2 weeks after the injection of the influenza vaccine.
  Other Names: Pneumovax NP® and Fluvic HA syringe®
  Arms: Sequential administration group

SUMMARY:
The immunogenicity of simultaneous administration of quadrivalent influenza vaccine and pneumococcal vaccine was unknown. The purpose of present study is to compare the immunogenicity of simultaneous administration of influenza vaccine and pneumococcal vaccine with that of separate administration.

DETAILED DESCRIPTION:
The immunogenicity of simultaneous administration of quadrivalent influenza vaccine and pneumococcal vaccine was unknown. We compare the immunogenicity of simultaneous administration of quadrivalent influenza vaccine and pneumococcal vaccine with that of separate administration.

162 Participants are randomly assigned to one of the two study groups; Simultaneous administration group: receive injections of pneumococcal vaccine and influenza vaccine simultaneously.

Sequential administration group: receive injections of pneumococcal vaccine 2 weeks after the injection of the influenza vaccine.

We compare the immunogenicity of the two groups.

ELIGIBILITY:
Inclusion Criteria:

* adults aged ≧65 years who had never received pneumococcal vaccine and quadrivalent influenza vaccine of 2015/2016 season

Exclusion Criteria:

* a sensitivity to pneumococcal and influenza vaccine
* received other inactivated vaccine within 14 days
* received other live vaccine within 28 days
* the presence of conditions known to impair pneumococcal vaccine response
* having malignant disease
* taking oral corticosteroids or immunosuppressive agent
* history of splenectomy
* history of an acute febrile illness or signs of severe acute illness at the time of vaccination
* other inappropriate condition to receive vaccination
* suffering an acute illness requiring antibiotics or steroids within the past month
* not expected to survive 12 months were also excluded

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 162 (Actual)
Dates: Start 2015-11; Primary Completion 2016-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kei Nakashima, MD, Principal Investigator — Department of Pulmonary Medicine, Kameda Medical Center
Locations (1):
- Department of Pulmonary Medicine, Kameda Medical Center, Kamogawa, Chiba, Japan

REFERENCES:
- [Background] Walter ND, Taylor TH, Shay DK, Thompson WW, Brammer L, Dowell SF, Moore MR; Active Bacterial Core Surveillance Team. Influenza circulation and the burden of invasive pneumococcal pneumonia during a non-pandemic period in the United States. Clin Infect Dis. 2010 Jan 15;50(2):175-83. doi: 10.1086/649208. PMID 20014948
- [Background] Oishi K, Yoshimine H, Watanabe H, Watanabe K, Tanimura S, Kawakami K, Iwagaki A, Nagai H, Goto H, Kudoh S, Kuriyama T, Fukuchi Y, Matsushima T, Shimada K, Matsumoto K, Nagatake T. Drug-resistant genes and serotypes of pneumococcal strains of community-acquired pneumonia among adults in Japan. Respirology. 2006 Jul;11(4):429-36. doi: 10.1111/j.1440-1843.2006.00867.x. PMID 16771912
- [Background] Hirst GK. THE QUANTITATIVE DETERMINATION OF INFLUENZA VIRUS AND ANTIBODIES BY MEANS OF RED CELL AGGLUTINATION. J Exp Med. 1942 Jan 1;75(1):49-64. doi: 10.1084/jem.75.1.49. PMID 19871167
- [Background] Dransfield MT, Nahm MH, Han MK, Harnden S, Criner GJ, Martinez FJ, Scanlon PD, Woodruff PG, Washko GR, Connett JE, Anthonisen NR, Bailey WC; COPD Clinical Research Network. Superior immune response to protein-conjugate versus free pneumococcal polysaccharide vaccine in chronic obstructive pulmonary disease. Am J Respir Crit Care Med. 2009 Sep 15;180(6):499-505. doi: 10.1164/rccm.200903-0488OC. Epub 2009 Jun 25. PMID 19556517
- [Background] Grabowska K, Hogberg L, Penttinen P, Svensson A, Ekdahl K. Occurrence of invasive pneumococcal disease and number of excess cases due to influenza. BMC Infect Dis. 2006 Mar 20;6:58. doi: 10.1186/1471-2334-6-58. PMID 16549029
- [Derived] Nakashima K, Aoshima M, Ohfuji S, Yamawaki S, Nemoto M, Hasegawa S, Noma S, Misawa M, Hosokawa N, Yaegashi M, Otsuka Y. Immunogenicity of simultaneous versus sequential administration of a 23-valent pneumococcal polysaccharide vaccine and a quadrivalent influenza vaccine in older individuals: A randomized, open-label, non-inferiority trial. Hum Vaccin Immunother. 2018;14(8):1923-1930. doi: 10.1080/21645515.2018.1455476. Epub 2018 May 14. PMID 29561248

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Started | 81 | 81
Completed | 81 | 76
Not Completed | 0 | 5

BASELINE CHARACTERISTICS:
Population: In the sequential administration group, we have 1 patient with eligibility error. Thus, we evaluated 81 patients in simultaneous administration group and 80 patients in sequential administration group after excluding 1 patient for ineligibility.
Groups:
- Total: Total of all reporting groups
Arm/Group | Simultaneous Administration Group | Sequential Administration Group | Total
Number analyzed (Participants) | 81 | 80 | 161
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.0 (5.1) | 70.2 (4.1) | 70.6 (4.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 33 | 31 | 64
  Male | 48 | 49 | 97

OUTCOME MEASURES:

1. Primary Outcome: The Number of Patients With Positive Antibody Response in Serotype 23F of Pneumococcal Antibody.
Description: The primary endpoint was the number of patients with positive antibody responses (≥2-fold increase in IgG concentrations 4-6 weeks after PPSV23 vaccination) in serotype 23F of the pneumococcal antibody.
Time Frame: 1month after the dose of PPV23
Population: In the sequential group, 5 patients were excluded from primary analysis because of the reasons below.
  1 patient: eligibility error, 1 patient: lost to follow-up (patient's decision), 3 patient: discontinued intervention (1 patient: fever, 2 patients: patient's decision
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Number analyzed (Participants) | 81 | 76
Participants | 63 | 59

2. Secondary Outcome: The Number of Patients With Positive Antibody Response in Serotype 3, 4, 6B, 1 4 and 19A of Pneumococcal Antibody.
Description: Positive antibody response was defined as ≥2-fold increase in IgG concentrations 4-6 weeks after PPSV23 vaccination in respective serotypes of the pneumococcal antibody.
Time Frame: 4 to 6 weeks after vaccination (P1), 24 weeks to 27 weeks after vaccination (P2)
Population: Immunogenicity was assessed in patients who received the allocated intervention (i.e., received at least 1 dose of the study vaccine), and had a blood sample taken within the planned time period.intervention (1 patient: fever, 2 patients: patient's decision
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Number analyzed (Participants) | 81 | 76
Participants
  4-6 weeks after vaccination 3 | 56 | 52
  4-6 weeks after vaccination 4 | 54 | 66
  4-6 weeks after vaccination 6B | 59 | 63
  4-6 weeks after vaccination 14 | 49 | 67
  4-6 weeks after vaccination 19A | 61 | 59
  24-27 weeks after vaccination 3: number analyzed (Participants) | 81 | 72
  24-27 weeks after vaccination 3 | 59 | 51
  24-27 weeks after vaccination 4: number analyzed (Participants) | 81 | 72
  24-27 weeks after vaccination 4 | 58 | 67
  24-27 weeks after vaccination 6B: number analyzed (Participants) | 81 | 72
  24-27 weeks after vaccination 6B | 66 | 63
  24-27 weeks after vaccination 14: number analyzed (Participants) | 81 | 73
  24-27 weeks after vaccination 14 | 59 | 66
  24-27 weeks after vaccination 19A: number analyzed (Participants) | 81 | 73
  24-27 weeks after vaccination 19A | 67 | 63

3. Secondary Outcome: The Geometric Mean Concentrations of Specific Antibodies to the 6 Serotypes (23F, 3, 4, 6B 14 and 19A)
Description: Pneumococcal IgG concentrations were converted using natural log transformations and presented as a geometric mean concentration.
Time Frame: Before vaccination (at baseline; in designated P0), 4 to 6 weeks after vaccination (P1), 24 weeks to 27 weeks after vaccination (P2)
Population: Immunogenicity was assessed in patients who received the allocated intervention (i.e., received at least 1 dose of the study vaccine), and had a blood sample taken within the planned time period.
Measure: Geometric Mean (95% Confidence Interval); unit: micrograms per milliliter
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Number analyzed (Participants) | 81 | 76
micrograms per milliliter
  Before vaccination 23F | 0.40 [0.30 to 0.55] | 0.20 [0.15 to 0.26]
  Before vaccination 3 | 0.07 [0.06 to 0.09] | 0.07 [0.06 to 0.08]
  Before vaccination 4 | 0.08 [0.06 to 0.10] | 0.05 [0.04 to 0.06]
  Before vaccination 6B | 0.24 [0.18 to 0.31] | 0.14 [0.11 to 0.18]
  Before vaccination 14 | 0.68 [0.50 to 0.92] | 0.42 [0.32 to 0.57]
  Before vaccination 19A | 0.72 [0.55 to 0.94] | 0.49 [0.38 to 0.64]
  4-6 weeks after vaccination 23F | 2.04 [1.42 to 2.94] | 1.41 [0.98 to 2.04]
  4-6 weeks after vaccination 3 | 0.24 [0.19 to 0.31] | 0.21 [0.17 to 0.27]
  4-6 weeks after vaccination 4 | 0.24 [0.18 to 0.33] | 0.28 [0.20 to 0.39]
  4-6 weeks after vaccination 6B | 0.96 [0.69 to 1.32] | 0.96 [0.67 to 1.37]
  4-6 weeks after vaccination 14 | 2.78 [1.84 to 4.19] | 4.72 [3.14 to 7.09]
  4-6 weeks after vaccination 19A | 3.74 [2.69 to 5.19] | 2.92 [1.98 to 4.23]
  24-27 weeks after vaccination 23F | 2.12 [1.58 to 2.86] | 1.70 [1.18 to 2.46]
  24-27 weeks after vaccination 3 | 0.26 [0.21 to 0.34] | 0.24 [0.19 to 0.31]
  24-27 weeks after vaccination 4 | 0.30 [0.22 to 0.41] | 0.36 [0.27 to 0.48]
  24-27 weeks after vaccination 6B | 1.18 [0.88 to 1.57] | 1.29 [0.91 to 1.82]
  24-27 weeks after vaccination 14 | 3.57 [2.42 to 5.27] | 6.21 [4.23 to 9.13]
  24-27 weeks after vaccination 19A | 4.61 [3.47 to 6.11] | 3.38 [2.47 to 4.63]

4. Secondary Outcome: The Number of Patients With Seroprotection Rate in Quadrivalent Influenza Vaccine.
Description: Seroprotection rates (post-vaccination titer ≥1:40) were calculated to assess the immunogenicity of influenza vaccination.
Time Frame: 4 to 6 weeks after vaccination (I1) and 24 weeks to 27 weeks after vaccination (I2)
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Number analyzed (Participants) | 81 | 77
Participants
  4 to 6 weeks after vaccination : H1N1 | 68 | 60
  4 to 6 weeks after vaccination : H3N2 | 66 | 68
  4 to 6 weeks after vaccination : B texas | 33 | 45
  4 to 6 weeks after vaccination : B Phuket | 49 | 48
  24 weeks to 27 weeks after vaccination : H1N1: number analyzed (Participants) | 81 | 73
  24 weeks to 27 weeks after vaccination : H1N1 | 41 | 46
  24 weeks to 27 weeks after vaccination : H3N2: number analyzed (Participants) | 81 | 73
  24 weeks to 27 weeks after vaccination : H3N2 | 47 | 44
  24 weeks to 27 weeks after vaccination : B texas: number analyzed (Participants) | 81 | 73
  24 weeks to 27 weeks after vaccination : B texas | 18 | 11
  24 weeks to 27 weeks after vaccination : B Phuket: number analyzed (Participants) | 81 | 73
  24 weeks to 27 weeks after vaccination : B Phuket | 24 | 16

ADVERSE EVENTS:
Time Frame: Local reactions at the injection site as well as systemic reactions were monitored for 28 days in the group that received the simultaneous administration, and for 14 days after each injection in the sequential group.
Description: The population in which safety was assessed consisted of participants who received a minimum of 1 dose of the vaccine.
  In the sequential group, 2 patients were excluded from the evaluation of adverse events because of the reasons below.1 patient: eligibility error, 1 patient: discontinued intervention (patient's decision) Regarding pain of axilla (evaluated only patients who received pneumococcal vaccine), additional 2 patients were excluded because they did not receive pneumococcal vaccine.
Arm/Group | Simultaneous Administration Group | Sequential Administration Group
Serious Adverse Events (participants affected / at risk) | 0/81 | 0/80
Other Adverse Events (participants affected / at risk) | 20/81 | 31/79
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Simultaneous Administration Group (N=81) | Sequential Administration Group (N=79)
Fatigue (General disorders) | 9 | 19
Joint pain (Skin and subcutaneous tissue disorders) | 11 | 11
Pain of axilla (Skin and subcutaneous tissue disorders) | 4 | 4/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No